CLINICAL TRIAL: NCT04516824
Title: Experience of Workforce From Orthopaedic and Spine Center Ghurki Trust Hospital Pakistan During COVID-19
Brief Title: Experience of Orthopaedic and Spine Center Pakistan During COVID-19
Status: Completed | Type: Observational
Sponsor: Ghurki Trust and Teaching Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 30
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Orthopaedic Disorders
Keywords: COVID 19; Orthopaedic conditions; Orthopaedic Surgeries; Pakistan
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma,Spine cases,Arthroplasty,Arthroscopy, Miscellaneous
  Interventions: Procedure: Orthopaedic Surgical Procedures

INTERVENTIONS:
Procedure: Orthopaedic Surgical Procedures — Intramedullary nails, Dynamic Compression Plate, Dynamic Hip Screw, Manipulation Under Anaesthesia POP, Ilizarov, Cannulated Screw Fixators, Bipolar Hemiarthroplasty, Locking Compression Plate, AO External fixators, Tension Band Wiring Patella, Pelvis and Acetabulum Fixations, Elbow Reconstructions, K wiring, Disc Excision, Spine Fracture i-e TPSF, Posterior Cervical Decompression and LMS, Dura repair, AD cage,Bilateral Total Hip Replacement, Unilateral Total Hip Replacement, Bilateral Total Knee Replacement, Unilateral Total Knee Replacement, Knee Arthroscopy for Mensicectomy, Arthroscopic Anterior Cruciate Ligament reconstruction,Removal of Implant, Amputations, VAC dressings,Wound wash, Arthrotomy for Septic Arthritis, Biopsy

SUMMARY:
After the frightful outbreak in the city of Wuhan, China and its evidence of being contagious, governments around the world particularly United States in an effort to stop the transmission- imposed travel restrictions to and from China. Though it's a novel virus and little is known about it, the spread was drastic across the world. In fact the spread was so rapid that by end of February 2020, the number of new cases outside China had leveled up to 13 fold as compared to the number of cases in China. Moreover, the number of infected countries with COVID-19 tripled. The first two reported cases in Pakistan were from Karachi and Islamabad on 27 February 2020. These two cases presented with a recent travel history from Iran. The current statistics showed the confirmed cases in Pakistan reached upto 284,121 till 9 August 2020.

During the lockdown period most of the public hospitals and trust closed their Outpatient departments and started to deal with emergency cases only. However even in such situation there are some trust hospitals worth mentioning who never closed their services and worked day and night to entertain their patients by observing all the precautions and safety measures. Ghurki trust teaching hospital is one of them. This hospital adopted a SMART STRATEGY or SMART hospital lockdown.

Since 19th March 2020 till 13th July 2020, the period of lockdown, two thousand one hundred and sixty surgeries were performed by the orthopaedic team of Ghurki hospital. The breakup of surgeries during lockdown was as follows: 1514 cases of trauma, 173 procedures of spine, 51 for arthroplasty, 51 for arthroscopy, 21 for tumors and 350 miscellaneous. The team was available 24 hours, 7 days a week under the supervisor of Professor Amer Aziz, to play their part in these terrible circumstances.

DETAILED DESCRIPTION:
After the frightful outbreak in the city of Wuhan, China and its evidence of being contagious, governments around the world particularly United States in an effort to stop the transmission- imposed travel restrictions to and from China. Though it's a novel virus and little is known about it, the spread was drastic across the world. In fact the spread was so rapid that by end of February 2020, the number of new cases outside China had levelled up to 13 fold as compared to the number of cases in China. Moreover, the number of infected countries with COVID-19 tripled. The first two reported cases in Pakistan were from Karachi and Islamabad on 27 February 2020. These two cases presented with a recent travel history from Iran. The current statistics showed the confirmed cases in Pakistan reached upto 284,121 till 9 August 2020.

Regarding the Pakistan's government response to COVID-19, quick steps were taken to curtail the transmission of virus as China is in northeast of Pakistan and also shares its borders with Iran where the number of cases are increasing exceptionally. As an initial response Pakistan closed its borders with China and implies strict methods at the Pakistan-Iran border. Still, in the initial days of pandemic Pakistan lacked the diagnosis kits and relied on China and Japan for testing purpose. However, later Pakistan was able to receive kits and started testing samples.

Pakistan's federal government along with the Ministry of Health (Moh) initiated a plan known as "National Action Plan for Corona Virus Disease Pakistan". The basic motive behind developing this plan was to generate policies and methods to combat with the deadly virus across Pakistan. MoH managed to deliver crucial supplies like masks, gloves and suits to the doctors and paramedical staffs working at frontlines. A state of confusion existed at different levels in health care system in Pakistan, particularly in Orthopaedic departments of hospital where elective and emergency services were severely affected during the lockdown period that started from 19 March 2020.

Orthopaedic and Spine Center Ghurki Trust Teaching Hospital Lahore:

During the lockdown period most of the public hospitals and trust closed their Outpatient departments and started to deal with emergency cases only. Even the private hospitals were reluctant to perform elective and emergency orthopaedic procedures. This attitude was may be due to the information published from other countries on the post operative complications and reduction of orthopaedic procedures during the period. The closure of orthopaedic health services brings a great shock to poor people for whom trusts and foundations is the last hope as they cannot afford the private setups for their health care facilities. However even in such situation there are some trust hospitals worth mentioning who never closed their services and worked day and night to entertain their patients by observing all the precautions and safety measures. Ghurki trust teaching hospital is one of them. This hospital adopted a SMART STRATEGY or SMART hospital lockdown. The orthopaedic department divided the members into five teams performing a 1:5 rotations. Each team comprised of one professor, one assistant professor, one senior registrar and ten trainee residents. Similarly the other departments like anesthesia, paramedics, nurses and physiotherapists were also subdivided. Out of two hundred staff, thirty were tested positive for COVID-19 but they all were managed and returned to normal after home quarantine.

Orthopaedic Surgeries during COVID-19:

Since 19th March 2020 till 13th July 2020, the period of lockdown, two thousand one hundred and sixty surgeries were performed by the orthopaedic team of Ghurki hospital. The breakup of surgeries during lockdown was as follows: 1514 cases of trauma, 173 procedures of spine, 51 for arthroplasty, 51 for arthroscopy, 21 for tumors and 350 miscellaneous. The team was available 24 hours, 7 days a week under the supervisor of Professor Amer Aziz, to play their part in these terrible circumstances. The team started their day with recitation of Quranic prayer which is translated as "In the name of Allah by whose name harm cannot be done by anything in the earth or in heavens. He is All-Hearing, All-Seeing" (Tirmidhi, Hadith: 3388). The smart approach utilized was that the patients were operated as soon as possible preferably within first twenty four hours and discharged them early also one to two days post op in most cases with complete education. All the patients were screened for COVID but Polymerase Chain Reaction test (PCR) and Pulmonary High-Resolution Computed Tomography (HRCT) was not done in all the patients unless if they presented with suspicious history. Fortunately, none of the patient tested positive pre operatively. Strict asepsis was observed during the period.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for surgical procedure
* Less affording patients coming from remote areas with the need of immediate orthopaedic surgery
* Urgent elective and emergency procedures

Exclusion Criteria:

* Elective surgery cases which were not urgent
* Patients in whom conservative management could be considered.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient ≥ 18 years old in which urgent elective and emergency orthopaedic surgical procedures were needed during COVID-19 lock down period in Pakistan.
Sampling Method: Non-Probability Sample
Enrollment: 2160 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Clinical and functional characteristics | [Through study period, average 3 months]
  Describe the clinical and functional level of patients after surgery, hospitalized during lockdown period in our hospital

SECONDARY OUTCOMES:
Patient's journey | [Through study period, average 3 months]
  Describe patient's experience during the period of lockdown in our center

CONTACTS AND LOCATIONS:
Overall Officials: Prof Amer Aziz, Study Director — Orthopaedic and Spine Center Ghurki Trust Hospital Lahore Pakistan; Prof. Atiq Uz Zaman, Study Chair — Orthopaedic and Spine Center Ghurki Trust Hospital Lahore Pakistan; Prof Rizwan Akram, Study Chair — Orthopaedic and Spine Center Ghurki Trust Hospital Lahore Pakistan; Prof. Ijaz Ahmad, Study Chair — Orthopaedic and Spine Center Ghurki Trust Hospital Lahore Pakistan; Dr. Ashfaq Jadoon, Study Chair — Orthopaedic and Spine Center Ghurki Trust Hospital Lahore Pakistan; Dr. Majid Cheema, Study Chair — Orthopaedic and Spine Center Ghurki Trust Hospital Lahore Pakistan; Dr. Samreen Sadiq, Study Chair — Lahore College of Physical Therapy LMDC GTTH
Locations (1):
- Ghurki trust hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No